CLINICAL TRIAL: NCT00668148
Title: A Five-Tier, Phase 2 Open-Label Study of IMC-A12 Administered as a Single Agent Every 2 Weeks in Patients With Previously-Treated, Advanced or Metastatic Soft Tissue and Ewing's Sarcoma/PNET
Brief Title: A Five-Tier, Open-Label Study of IMC-A12 in Advanced Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13925; 2007-006719-21 (EudraCT Number); CP13-0707 (Other: ImClone, LLC); I5A-IE-JAEC (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Ewing's Sarcoma /Peripheral Neuroectodermal Tumor (PNET); Rhabdomyosarcoma; Leiomyosarcoma; Adipocytic Sarcoma; Synovial Sarcoma
Keywords: Sarcoma; Ewing's sarcoma / peripheral neuroectodermal tumor (PNET);; rhabdomyosarcoma;; leiomyosarcoma;; adipocytic sarcoma; synovial sarcoma
MeSH Terms: conditions — Rhabdomyosarcoma; Leiomyosarcoma; Sarcoma, Synovial; Sarcoma; Sarcoma, Ewing; Neuroectodermal Tumors, Primitive, Peripheral; Neuroectodermal Tumors, Primitive | interventions — cixutumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMC-A12 (cixutumumab) (Experimental)
  Interventions: Biological: IMC-A12 (cixutumumab)

INTERVENTIONS:
Biological: IMC-A12 (cixutumumab) — Ewing's Sarcoma/PNET
  10 milligrams per kilogram (mg/kg) intravenous (IV) infusion every two weeks.
  A treatment cycle will be defined as 6 weeks, with radiological evaluation at every cycle.
  Other Names: cixutumumab; LY3012217
Biological: IMC-A12 (cixutumumab) — Rhabdomyosarcoma
  10 mg/kg IV infusion every two weeks.
  A treatment cycle will be defined as 6 weeks, with radiological evaluation at every cycle.
  Other Names: cixutumumab; LY3012217
Biological: IMC-A12 (cixutumumab) — Leiomyosarcoma
  10 mg/kg IV infusion every two weeks.
  A treatment cycle will be defined as 6 weeks, with radiological evaluation at every cycle.
  Other Names: cixutumumab; LY3012217
Biological: IMC-A12 (cixutumumab) — Adipocytic sarcoma
  10 mg/kg IV infusion every two weeks.
  A treatment cycle will be defined as 6 weeks, with radiological evaluation at every cycle.
  Other Names: cixutumumab; LY3012217
Biological: IMC-A12 (cixutumumab) — Synovial sarcoma
  10 mg/kg IV infusion every two weeks.
  A treatment cycle will be defined as 6 weeks, with radiological evaluation at every cycle.
  Other Names: cixutumumab; LY3012217

SUMMARY:
This multicenter study will enroll approximately 185 participants with metastatic or advanced sarcoma, to assess the effectiveness and safety of IMC-A12 monotherapy for this indication. Participants will be stratified into five tiers according to diagnosis:

1. Ewing's sarcoma/peripheral neuroectodermal tumor (PNET)
2. rhabdomyosarcoma
3. leiomyosarcoma
4. adipocytic sarcoma
5. synovial sarcoma.

A total of 85 participants will be enrolled initially, 17 in each tier. Participants will receive single agent IMC-A12 every 2 weeks. A treatment cycle will be defined as 6 weeks, with radiological evaluation at every cycle.

Safety and response in the initial 17 participants in each tier will be used to determine whether to extend enrollment to the target total of 37 participants per tier.

DETAILED DESCRIPTION:
The purpose of this study is to determine the progression-free survival (PFS) rate assessed 12 weeks after the initiation of IMC-A12 monotherapy, administered every 2 weeks to participants with previously-treated, advanced or metastatic soft tissue and Ewing's sarcoma/PNET.

ELIGIBILITY:
Inclusion:

* Histologically or cytologically-confirmed sarcoma of one of the following histologies: (1) Ewing's sarcoma / PNET; (2) rhabdomyosarcoma; (3) leiomyosarcoma; (4) adipocytic sarcoma; or (5) synovial sarcoma
* Has measurable disease, at least one lesion ≥ 2 centimeters (cm) on conventional measurement techniques or ≥ 1 cm on spiral computed tomography (CT) scan
* Has at least one measurable lesion located outside of a previously irradiated area
* Has radiographic documentation of disease progression within 6 months prior to study entry
* Has relapsed, refractory, and/or metastatic disease, incurable by surgery, radiotherapy, or other conventional systemic therapy
* Been considered ineligible for systemic chemotherapy or received at least one previous regimen for relapsed, refractory, and/or metastatic disease
* Adequate hematologic function
* Has adequate hepatic function
* Has adequate coagulation function
* Has adequate renal function
* Has fasting serum glucose < 120 milligrams per deciliter (mg/dL) or below the upper limit of normal (ULN)
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation

Exclusion:

* Has uncontrolled brain or leptomeningeal metastases
* Not recovered to grade ≤ 1 from adverse events due to agents administered more than 3 weeks prior to study entry
* Is receiving any other investigational agent(s)
* Major surgery, hormonal therapy (other than replacement), chemotherapy, radiotherapy, or any form of investigational therapy within 3 weeks prior to enrollment
* History of treatment with other agents targeting the insulin-like growth factor-I receptor (IGF-IR)
* History of allergic reactions attributed to compounds of chemical or biologic composition similar to that of IMC-A12
* Has poorly controlled diabetes mellitus
* Is receiving therapy with immunosuppressive agents
* Is pregnant or breastfeeding

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2008-07; Primary Completion 2010-10 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E-mail: ClinicalTrials@ ImClone.com, Study Director — Eli Lilly and Company
Locations (18):
- United States (6):
  - ImClone Investigational Site, Aurora, Colorado
  - ImClone Investigational Site, Orlando, Florida
  - ImClone Investigational Site, Metairie, Louisiana
  - ImClone Investigational Site, Detroit, Michigan
  - ImClone Investigational Site, St Louis, Missouri
  - ImClone Investigational Site, Columbus, Ohio
- Belgium (3):
  - ImClone Investigational Site, Brussels
  - ImClone Investigational Site, Leuven
  - ImClone Investigational Site, Wilrijk
- France (4):
  - ImClone Investigational Site, Bordeaux
  - ImClone Investigational Site, Lyon
  - ImClone Investigational Site, Paris
  - ImClone Investigational Site, Toulouse
- Germany (2):
  - ImClone Investigational Site, Dresden
  - ImClone Investigational Site, Mannheim
- ImClone Investigational Site, Leiden, Netherlands
- ImClone Investigational Site, Warsaw, Poland
- ImClone Investigational Site, Barcelona, Spain

REFERENCES:
- [Derived] Asmane I, Watkin E, Alberti L, Duc A, Marec-Berard P, Ray-Coquard I, Cassier P, Decouvelaere AV, Ranchere D, Kurtz JE, Bergerat JP, Blay JY. Insulin-like growth factor type 1 receptor (IGF-1R) exclusive nuclear staining: a predictive biomarker for IGF-1R monoclonal antibody (Ab) therapy in sarcomas. Eur J Cancer. 2012 Nov;48(16):3027-35. doi: 10.1016/j.ejca.2012.05.009. Epub 2012 Jun 7. PMID 22682017

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Presented are the reasons the participants discontinued from study treatment.
Groups:
- Entire Study Population: IMC-A12 (cixutumumab) 10 milligrams per kilogram (mg/kg) dose administered as intravenous infusion over a period of 1 hour once every 2 weeks (6-week cycle). Participants were stratified into 5 arms according to the disease condition: Ewing's Sarcoma/peripheral neuroectodermal tumor (PNET), rhabdomyosarcoma, leiomyosarcoma, adipocytic sarcoma, and synovial sarcoma.
  Treatment was continued until there was evidence of disease progression, unacceptable toxicity, or withdrawal of consent.
Period: Overall Study
Arm/Group | Entire Study Population
Started | 113
Received at Least 1 Dose of Study Drug | 111
Completed | 103
Not Completed | 10
Not completed — Adverse Event | 5
Not completed — Subject Non-compliance | 1
Not completed — Progressive Disease Before Treatment | 2
Not completed — Withdrawal of Consent | 2

BASELINE CHARACTERISTICS:
Population: Enrolled participants who received at least 1 dose of study drug.
Groups:
- Entire Study Population: IMC-A12 (cixutumumab) 10 mg/kg dose administered as intravenous infusion over a period of 1 hour once every 2 weeks (6-week cycle). Participants were stratified into 5 arms according to the disease condition: Ewing's Sarcoma/PNET, rhabdomyosarcoma, leiomyosarcoma, adipocytic sarcoma, and synovial sarcoma.
  Treatment was continued until there was evidence of disease progression, unacceptable toxicity, or withdrawal of consent.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 111
Age, Continuous [Median (Full Range); unit: years] | 47.0 (10.3) [17 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 102
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 101
  Black | 5
  Other | 5
Region of Enrollment [Count of Participants; unit: Participants]
  France | 15
  United States | 50
  Poland | 7
  Spain | 9
  Belgium | 23
  Germany | 1
  Netherlands | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression-Free Survival (PFS) at 12 Weeks
Description: PFS at 12 weeks was reported by disease condition and defined as the percentage of participants who have neither experienced disease progression nor died at 12 weeks after the date of first dose. Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST, version 1.0) criteria. Progressive Disease (PD) was defined as having at least a 20% increase in sum of the longest diameter of target lesions or the appearance of new lesions. Percentage of participants is calculated as the total number of participants with PFS at 12 weeks divided by the total number of participants treated then multiplied by 100.
Time Frame: Baseline to Disease Progression or Death Due to Any Cause Up To 12 Weeks
Population: Enrolled participants who received any quantity of IMC-A12.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Ewing's Sarcoma/PNET; Rhabdomyosarcoma; Leiomyosarcoma; Adipocytic Sarcoma; Synovial Sarcoma: IMC-A12 (cixutumumab) 10 mg/kg dose administered as intravenous infusion over a period of 1 hour once every 2 weeks (6-week cycle). Treatment was continued until there was evidence of disease progression, unacceptable toxicity, or withdrawal of consent.
- Total: Total of all reporting groups.
Arm/Group | Ewing's Sarcoma/PNET | Rhabdomyosarcoma | Leiomyosarcoma | Adipocytic Sarcoma | Synovial Sarcoma | Total
Number analyzed (Participants) | 18 | 17 | 22 | 37 | 17 | 111
percentage of participants | 27.3 [8.5 to 50.4] | 12.5 [2.1 to 32.8] | 25.4 [8.4 to 46.8] | 50.0 [32.9 to 64.9] | 21.4 [5.2 to 44.8] | 31.9 [23.0 to 41.1]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was reported by disease condition and defined as the interval from the date of first dose until disease progression or death whichever occurred earlier. Response was defined using RECIST, version 1.0 criteria. PD was defined as having at least a 20% increase in sum of the longest diameter of target lesions or the appearance of new lesions. PFS was censored at the date of the last objective progression-free disease assessment for participants who did not experience disease progression or death.
Time Frame: Baseline to measured PD (up to 105.4 weeks)
Population: Enrolled participants who received any quantity of IMC-A12. Three (3) participants in Ewing's sarcoma/PNET, 1 participant in rhabdomyosarcoma, 4 participants in leiomyosarcoma, 6 participants in adipocytic sarcoma, and 3 participants in synovial sarcoma groups were censored for analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Ewing's Sarcoma/PNET; Rhabdomyosarcoma; Leiomyosarcoma; Adipocytic Sarcoma; Synovial Sarcoma: IMC-A12 (cixutumumab) 10 mg/kg dose administered as intravenous infusion over a period of 1 hour once every 2 weeks (6-week cycle). Treatment was continued until there was evidence of disease progression, unacceptable toxicity, or withdrawn consent.
Arm/Group | Ewing's Sarcoma/PNET | Rhabdomyosarcoma | Leiomyosarcoma | Adipocytic Sarcoma | Synovial Sarcoma | Total
Number analyzed (Participants) | 18 | 17 | 22 | 37 | 17 | 111
weeks | 6.4 [5.1 to 12.1] | 6.1 [5.1 to 7.3] | 6.0 [5.4 to 11.0] | 12.1 [6.0 to 17.7] | 6.4 [5.6 to 11.9] | 6.7 [6.0 to 11.0]

3. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) [Objective Response Rate (ORR)]
Description: ORR was reported by disease condition and defined as the percentage of participants achieving either CR or PR. Response was defined using RECIST, version 1.0 criteria. CR was defined as the disappearance of all target lesions. PR was defined as having at least a 30% decrease in sum of longest diameter of target lesions. Percentage of participants is calculated as a total number of participants with CR or PR divided by the total number of participants treated then multiplied by 100.
Time Frame: Baseline to measured PD (up to 105.4 weeks)
Population: Enrolled participants who received any quantity of IMC-A12.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ewing's Sarcoma/PNET | Rhabdomyosarcoma | Leiomyosarcoma | Adipocytic Sarcoma | Synovial Sarcoma | Total
Number analyzed (Participants) | 18 | 17 | 22 | 37 | 17 | 111
percentage of participants | 5.6 [0.1 to 27.3] | 0 [0.0 to 19.5] | 0 [0.0 to 15.4] | 2.7 [0.1 to 14.2] | 0 [0.0 to 19.5] | 1.8 [0.2 to 6.4]

4. Secondary Outcome: Time to Response
Time Frame: Baseline to first evidence of confirmed CR or PR (up to 105.4 weeks)
Population: Zero participants analyzed. Time to Response for CR and PR data was not collected for analysis per study report.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 0

5. Secondary Outcome: Duration of Response
Time Frame: Date of first response to the date of progression or death due to any cause (up to 105.4 weeks)
Population: Zero participants analyzed. Duration to Response for CR and PR data was not collected for analysis per study report.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival (OS)
Description: OS was reported by disease condition and defined as the duration from the date of enrollment to the date of death from any cause. For participants who were alive, OS was censored at the date of last follow-up visit or at the date of last contact.
Time Frame: Baseline to date of death from any cause (up to 112.9 weeks)
Population: Enrolled participants who received any quantity of IMC-A12. Five (5) participants in Ewing's sarcoma/PNET, 4 participants in rhabdomyosarcoma, 12 participants in leiomyosarcoma, 11 participants in adipocytic sarcoma, and 5 participants in synovial sarcoma groups were censored for analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Ewing's Sarcoma/PNET | Rhabdomyosarcoma | Leiomyosarcoma | Adipocytic Sarcoma | Synovial Sarcoma | Total
Number analyzed (Participants) | 18 | 17 | 22 | 37 | 17 | 111
weeks | 24.1 [12.6 to 37.6] | 23.6 [8.9 to 52.1] | NA [25.7 to NA] — Median OS and upper limit of 95% confidence interval could not be mathematically calculated due to high censoring rate. | 46.4 [31.3 to 61.1] | 56.3 [22.3 to 71.3] | 38.4 [31.1 to 52.0]

7. Secondary Outcome: Percentage of Participants With Best Overall Response [Clinical Benefit Rate (CBR)]
Description: CBR was reported by disease condition. Response was defined using RECIST, version 1.0 criteria. CR was defined as the disappearance of all target lesions. PR was defined as having at least a 30% decrease in sum of longest diameter of target lesions. Stable Disease (SD) was defined as small changes that did not meet the above criteria. Percentage of participants with best overall response is calculated as a total number of participants with CR or PR or SD divided by the total number of participants treated then multiplied by 100.
Time Frame: Baseline through study completion (up to 105.4 weeks)
Population: Enrolled participants who received any quantity of IMC-A12.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ewing's Sarcoma/PNET | Rhabdomyosarcoma | Leiomyosarcoma | Adipocytic Sarcoma | Synovial Sarcoma | Total
Number analyzed (Participants) | 18 | 17 | 22 | 37 | 17 | 111
percentage of participants | 33.3 [13.3 to 59.0] | 23.5 [6.8 to 49.9] | 40.9 [20.7 to 63.6] | 56.8 [39.5 to 72.9] | 35.3 [14.2 to 61.7] | 41.4 [32.2 to 51.2]

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) or Deaths
Description: TEAEs were defined as serious and other non-serious AEs that occurred or worsened after study treatment (regardless of causality). Data presented are the number of participants who experienced TEAEs, serious TEAEs, and deaths during the study including the 30-day follow-up. A summary of serious and other non-serious AEs regardless of causality is located in the Reported Adverse Event module.
Time Frame: Baseline through study completion (up to 112.9 weeks)
Population: Enrolled participants who received any quantity of IMC-A12.
Measure: Count of Participants; unit: Participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 111
Participants
  Any TEAE | 108
  Serious TEAE | 56
  Deaths Due to Disease Progression | 10
  Death Due to Other Cause | 1
  Death Due to AE | 1

9. Secondary Outcome: Serum Anti-IMC-A12 Antibody Assessment (Immunogenicity)
Time Frame: 30-day safety follow-up
Population: Zero participants analyzed. Analysis was not performed due to lack of available assay.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Entire Study Population
Serious Adverse Events (participants affected / at risk) | 56/111
Other Adverse Events (participants affected / at risk) | 97/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Entire Study Population (N=111)
Anaemia (Blood and lymphatic system disorders) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (2)
Chorioretinopathy (Eye disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Malabsorption (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Disease progression (General disorders) | 14 (16)
General physical health deterioration (General disorders) | 2 (2)
Infusion related reaction (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 6 (7)
Catheter related infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Endocarditis bacterial (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Pyelonephritis (Infections and infestations) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 3 (3)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/54 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Entire Study Population (N=111)
Anaemia (Blood and lymphatic system disorders) | 13 (29)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (10)
Abdominal pain (Gastrointestinal disorders) | 10 (24)
Constipation (Gastrointestinal disorders) | 16 (18)
Diarrhoea (Gastrointestinal disorders) | 25 (42)
Nausea (Gastrointestinal disorders) | 28 (32)
Vomiting (Gastrointestinal disorders) | 15 (18)
Asthenia (General disorders) | 17 (81)
Chest pain (General disorders) | 6 (6)
Fatigue (General disorders) | 26 (36)
Mucosal inflammation (General disorders) | 6 (7)
Oedema peripheral (General disorders) | 7 (8)
Activated partial thromboplastin time prolonged (Investigations) | 6 (7)
Alanine aminotransferase increased (Investigations) | 6 (8)
Blood creatinine increased (Investigations) | 13 (22)
Haemoglobin decreased (Investigations) | 6 (19)
Weight decreased (Investigations) | 11 (14)
Anorexia (Metabolism and nutrition disorders) | 19 (22)
Hyperglycaemia (Metabolism and nutrition disorders) | 22 (60)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (10)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 (20)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (8)
Dizziness (Nervous system disorders) | 6 (7)
Headache (Nervous system disorders) | 12 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (14)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.